CLINICAL TRIAL: NCT02982226
Title: A Comparative Study of Injectable Human Amniotic Allograft (ReNu™) Versus Corticosteroids for Plantar Fasciitis: A Prospective, Randomized, Blinded Study
Brief Title: ReNu™ vs. Corticosteroids for the Treatment of Plantar Fasciitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NuTech Medical, Inc (Industry)
Collaborators: MileStone Research Organization (Industry); Organogenesis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RD-2015-08-05
Record Dates: First submitted 2016-11-29; First posted 2016-12-05 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Fasciitis, Plantar
Keywords: Plantar Fasciitis; Jogger's Heel; ReNu
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ReNu Injection (Experimental): Plantar Fascia injection with ReNu. ReNu is an allograft tissue composed of particularized amniotic membrane and cell from the amniotic fluid.
  Interventions: Other: ReNu Injection
- Corticosteroid Injection (Active Comparator): Plantar Fascia injection with Corticosteroids.
  Interventions: Other: Corticosteroid Injection

INTERVENTIONS:
Other: ReNu Injection — ReNu is an allograft tissue composed of particularized amniotic membrane and cell from the amniotic fluid.
  Arms: ReNu Injection
Other: Corticosteroid Injection — Corticosteroids are considered a standard of care for treatment of Plantar Fasciitis
  Arms: Corticosteroid Injection

SUMMARY:
The objective of this clinical trial is to evaluate both the safety and efficacy of the ReNu™ injection on pain and inflammation in subjects diagnosed with plantar fasciitis as compared to a Corticosteroid Injection which is considered standard of care.

DETAILED DESCRIPTION:
This is a two (2) arm evaluation in 150 subjects with plantar fasciitis. Patients will be treated with ReNu™(study treatment) or Corticosteroids (control).

At each follow-up visit, concomitant medications and adverse events shall be collected from each subject, and each subject shall complete following questionnaires:

* AOFAS Ankle-Hindfoot Score (AOFAS-AHS)
* Visual Analog Score (VAS)
* Single Answer Numeric Evaluation (SANE)
* Subject Satisfaction Score (at the 6 Month Follow Ups ONLY)

The subjects will be assessed at Baseline (pre-injection) using these scales and again at all subsequent study follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 to 75 inclusive
2. BMI less than 40
3. Actively practicing a contraception method, abstinent, surgically sterile, or post-menopausal (defined as no menses for a minimum of 12 months)
4. Reporting heel pain of >6 on a verbally administered 1-10 pain scale where 1 is no pain and 10 is extreme pain
5. Diagnosed with plantar fasciitis in either foot
6. Completed a minimum of two months of conservative, non-injection treatment/therapies (i.e., activity modification, icing, NSAIDs, orthotics, physical therapy, etc.)

Exclusion Criteria

1. Prior surgery on the affected foot
2. Prior injection treatment for plantar fasciitis within the past 6 months with steroids or tissue engineered materials just in the site seeking treatment
3. Clinical signs and symptoms of infection of foot in question
4. Evidence of significant neurological disease of either foot
5. Non-ambulatory
6. Presence of comorbidities that can be confused with or can exacerbate the condition including, but not limited to the following:

   * Calcaneal stress fracture
   * Nerve entrapment syndrome, such as Baxter's Nerve Entrapment or Tarsal Tunnel Syndrome
   * Plantar Fascial rupture
   * Systemic disorders associated with enthesiopathy, i.e., Gout, Reiter's syndrome, rheumatoid arthritis, etc.
   * Achilles tendonitis
   * Fat Pad Atrophy
   * Fibromyalgia
   * Diabetic Neuropathy
7. Pregnant, pregnant within the past six (6) months, breast feeding and/or desire to become pregnant during the course of the study, as verified by urine pregnancy test within one week prior to injection.
8. Has taken NSAID medication within the past 14 days, or other pain medication in the past day
9. History of more than two (2) weeks treatment with immuno-suppressants, including systemic corticosteroids or cytotoxic chemotherapy within one month prior to initial screening, or has receive such medications during the screening period, or are anticipated to require such medications during the course of the study.
10. Taking any investigational drug(s) or therapeutic device(s) within 30 days preceding screening
11. History of radiation therapy of the affected foot
12. Known history of having Acquired Immunodeficiency Syndrome (AIDS) or HIV
13. Involved in a Worker's Compensation Claim of any kind
14. Unable to understand the objectives of the trial
15. Presence of any condition(s) which, in the opinion of the investigator, would compromise the subject's ability to complete this study
16. Having a known history of poor adherence with medical treatment.
17. Express an unwillingness to receive human allograft tissue

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Change in AOFAS score from baseline | 6 months

SECONDARY OUTCOMES:
Change in VAS pain score from baseline | 6 months
Change in SANE function score from baseline | 6 months
Return to Normal Function between treatment groups | 6 months
  Assessed using questionnaire by the Principal Investigator (PI)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Ng, DPM, FACFAS, Principal Investigator — Advanced Orthopedics
Locations (6):
- United States (6):
  - Advanced Orthopedics, Denver, Colorado
  - Orlando Food and Ankle Clinic, Orlando, Florida
  - The Iowa Clinic Foot and Ankle Surgery, West Des Moines, Iowa
  - Lower Extremity Institute of Research & Therapy (LEIRT), Poland, Ohio
  - Geisinger, Danville, Pennsylvania
  - The Vancouvover Clinic, Vancouver, Washington

IPD SHARING:
Plan to Share IPD: No